CLINICAL TRIAL: NCT04093375
Title: Primary Radical Prostatectomy Versus Primary Radiotherapy for Locally Advanced Prostate Cancer: an Open Randomized Clinical Trial
Brief Title: Radical Prostatectomy Versus Radical Radiotherapy for Locally Advanced Prostate Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Changhai Hospital (Other); Zhejiang University (Other); Sun Yat-sen University (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019CR101
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-05

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radical Prostatectomy (Experimental): Patients with locally advanced prostate adenocarcinoma receives Radical Prostatectomy with or without enlarged lymph node dissection
  Interventions: Procedure: Radical Prostatectomy
- Radical Radiotherapy (Active Comparator): Patients with locally advanced prostate adenocarcinoma receives Radical Radiotherapy with adjuvant androgen deprivation therapy
  Interventions: Other: Radical Radiotherapy

INTERVENTIONS:
Procedure: Radical Prostatectomy — Radical prostatectomy with or without androgen deprivation therapy
  Arms: Radical Prostatectomy
Other: Radical Radiotherapy — Radical Radiotherapy with adjuvant androgen deprivation therapy
  Arms: Radical Radiotherapy

SUMMARY:
This prospective, open randomized clinical trial seeks to investigate whether radical prostatectomy with androgen deprivation therapy improves prostate-cancer specific survival and quality of life in comparison with radical radiation treatment with androgen deprivation therapy among patients diagnosed locally advanced prostate cancer. Lack of extensive PSA screening in mainland China, many new cases of prostate cancer are LAPCa. Surgery and/or radiation plus attempted chemotherapy are curative treatment for advanced solid malign tumors to control and eliminate the local and micro metastases. LAPCa is easy to metastasis, relapse and has a poor prognosis. For LAPCa, a single RP approach is generally not the preferred option because it is generally considered that radical surgery is difficult to completely remove the lesion and the long-term prognosis is not ideal. However, androgen deprivation therapy promotes the prognosis of LAPCa with lymph nodes or seminal vesicle metastases and improves the local control rate of tumor. What is more, for early localized prostate cancer, RT has similar efficacy to RP, for advanced tumor RT can not only relieve urinary tract obstruction and other symptoms, but also improve biochemical progression free survival and local oncological control. A randomized clinical trial comparing two multimodal treatment including RP or RT with ADT regimens is therefore warranted.

ELIGIBILITY:
Inclusion Criteria:

1. 18≤Age ≤75, at the time of randomization.
2. Confirmed as non-metastatic prostate adenocarcinoma by transrectal ultrasound biopsy in six months before enrollment and untreated.
3. Tumor stage (T, M, N): according to 2018 NCCN prostate cancer guidelines T3 stage Significant extra-capsular tumor extension M0 (no sign of distant metastases) Nx (regional lymph nodes cannot be assessed). For patients with T4, the tumor should be confined to the bladder neck, and bilateral ureters should not be invaded.
4. WHO score 0-1, ECOG score 0-2, and ASA grade I-III.
5. At least 5 years life expectancy.
6. The general condition and mental status of patients shall permit observation in accordance with the study protocol.
7. Signed Informed consent.

Exclusion Criteria:

1. Concomitant with other malignancies.
2. With severe systemic disease (cardio-cerebrovascular disease, etc.) cannot tolerate surgery or radiotherapy.
3. Clinical significant abnormal laboratory values at the discretion of the investigator, e.g. severe kidney function GFR < 30 ml/ml or elevated liver transaminases above > 10 ULN.
4. Involved in other clinical trials simultaneously.
5. Any medical condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cause-specific survival | Up to 5 years
Overall survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhihua Wang, M.D ass. prof, Principal Investigator — Tongji Hospital

IPD SHARING:
Plan to Share IPD: No